CLINICAL TRIAL: NCT03946332
Title: Physical Exercises for Patient Undergoing Hematopoietic Stem Cell Transplantation for Multiple Myeloma: a Controlled Randomised Prospective Multicentre Longitudinal Study.
Brief Title: Physical Activity for Myeloma Autograft Longitudinal Study
Acronym: PAMAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: University Hospital, Rouen (Other); University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PI2018_843_0008
Record Dates: First submitted 2019-05-09; First posted 2019-05-10 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Physical Activity; Multiple Myeloma; Quality of Life
Keywords: physical activity; multiple myeloma; autologous stem cell transplantation; quality of life; physical conditioning
MeSH Terms: conditions — Motor Activity; Multiple Myeloma | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical exercise arm (Experimental): patients will benefit regularly from a physical exercises program during their hospitalization. When going back home, they will be given a practical help kit with specific equipment (dumbbell, elastic), an actimeter with heart rate monitoring (in order to have an objective collection of the physical practice in addition to a self-evaluation) and a physical exercises program on paper and video supports, that patients would have learnt during their hospitalization. Furthermore, SMS will be regularly sent to remind them to practice
  Interventions: Behavioral: Physical exercises
- controlled arm (Active Comparator): patients will be hospitalized in the same conditions than the experimental group and will be able to practice if they want.
  Interventions: Behavioral: Optional physical exercises

INTERVENTIONS:
Behavioral: Physical exercises — patients will benefit regularly from a physical exercises program during their hospitalization. When going back home, they will be given a practical help kit with specific equipment (dumbbell, elastic), an actimeter with heart rate monitoring (in order to have an objective collection of the physical practice in addition to a self-evaluation) and a physical exercises program on paper and video supports, that patients would have learnt during their hospitalization.
  Arms: Physical exercise arm
Behavioral: Optional physical exercises — patients will be proposed for the physical exercises and will practice them if they want.
  Arms: controlled arm

SUMMARY:
Physical exercises program is known to improve quality of life, chronical fatigue and appears to be a behavioural recommendation against cancer as primary and tertiary prevention. Nutritional status is also important in cancer patients: a loss of 5% of weight increases the complication risks and decreases survival and the quality of life. Interactions between physical activity and haematological malignancies are less described compared to solid cancers. Methodology and protocols are also heterogeneous. Supervised exercises program improves the physical condition and the quality of life; however there are few randomised studies versus a controlled group. Post autograft evaluation for myeloma patients showed a physical deficit with increased fat mass, but in this particular population physical exercises need to be more explored. This project is a randomised study versus controlled group that evaluates supervised physical exercises program in a homogenous population: patients under-65-years-old with multiple myeloma and who will undergo autologous stem cell transplantation.

DETAILED DESCRIPTION:
Physical exercises program is known to improve quality of life, chronical fatigue and appears to be a behavioural recommendation against cancer as primary and tertiary prevention. Nutritional status is also important in cancer patients: a loss of 5% of weight increases the complication risks and decreases survival and the quality of life. Interactions between physical activity and haematological malignancies are less described compared to solid cancers. This multicentre project is a randomised study versus controlled group that evaluates supervised physical exercises program in a homogenous population: patients under-65-years-old with multiple myeloma and who will undergo autologous stem cell transplantation. The hypothesis of this study is that a supervised physical exercises program during and after autograft might have a positive impact on the physical capacities and the quality of life.

In the experimental arm, patients will benefit regularly from a physical exercises program during their hospitalization. When going back home, they will be given a practical help kit with specific equipment (dumbbell, elastic), an actimeter with heart rate monitoring (in order to have an objective collection of the physical practice in addition to a self-evaluation) and a physical exercises program on paper and video supports, that patients would have learnt during their hospitalization. Furthermore, SMS will be regularly sent to remind them to practice. In the controlled arm, patients will be hospitalized in the same conditions than the experimental group and can practice if they want. At the end of the hospitalization, they will receive a paper document with global informations about physical exercises including a few simple exercises. Evaluations will be carried out in both arms at day 0, day 30 and day 90 from autograft. The post graft follow up will be done at the same time as the medical consultation and before the maintenance treatment.

ELIGIBILITY:
Inclusion Criteria:

* Under 65-year-old patient
* more than 18 years old
* Hospitalized for autologous stem cell transplantation
* First or second line therapy for multiple myeloma
* Chemotherapy regimen with melphalan
* Patient affiliated to the social security system
* Signed informed consent form
* Patient who have computer and internet connection at home

Exclusion Criteria:

* Over-65-year-old patient
* Other haematological malignancies
* More than 2 treatment lines
* Other regimen of chemotherapy for autograft than melphalan
* Contraindication to physical exercises: uncontrolled arterial hypertension or diabetes, heart or respiratory failure, psycho-cognitive disorders that may compromise the physical exercises program
* dialyzed patient
* Adult patient under tutelage

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2023-05-01 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Measure of quality of life with EORTC QLQ-C30 questionnaire | at day 0 from autograft as patient will be hospitalized.
  The quality of life will be measure with the EORTC quality QLQ-C30 questionnaire to assess the quality of life of cancer patients. Scales range in score is from 0 to 100. A high score for a functional scale represents a high/healthy level of functioning whereas a high score for a symptom scale or item represents a high level of symptomatology or problems.
Measure of quality of life with EORTC QLQ-C30 questionnaire | at day 30 from autograft as patient will be hospitalized.
  The quality of life will be measure with the EORTC quality QLQ-C30 questionnaire to assess the quality of life of cancer patients. Scales range in score is from 0 to 100. A high score for a functional scale represents a high/healthy level of functioning whereas a high score for a symptom scale or item represents a high level of symptomatology or problems.
Measure of quality of life with EORTC QLQ-C30 questionnaire | at day 90 from autograft as patient will be hospitalized.
  The quality of life will be measure with the EORTC quality QLQ-C30 questionnaire to assess the quality of life of cancer patients. Scales range in score is from 0 to 100. A high score for a functional scale represents a high/healthy level of functioning whereas a high score for a symptom scale or item represents a high level of symptomatology or problems.
Measure of quality of life with QLQ-MY20 questionnaire | at day 0 from autograft as patient will be hospitalized.
  The quality of life will be measure with the QLQ-MY20 questionnaire to assess the quality of life of cancer patients.
  QLQ-MY20 domain scores are averaged and transformed linearly to a score ranging from 0-100. A high score for Disease Symptoms and Side Effects of Treatment represents a high level of symptomatology or problems, whereas a high score for Future Perspective and Body Image represents better outcomes.
Measure of quality of life measured with QLQ-MY20 questionnaire | at day 30 from autograft as patient will be hospitalized.
  The quality of life will be measure with the QLQ-MY20 questionnaire to assess the quality of life of cancer patients.
  QLQ-MY20 domain scores are averaged and transformed linearly to a score ranging from 0-100. A high score for Disease Symptoms and Side Effects of Treatment represents a high level of symptomatology or problems, whereas a high score for Future Perspective and Body Image represents better outcomes.
Measure of quality of life measured with QLQ-MY20 questionnaire | at day 90 from autograft as patient will be hospitalized.
  The quality of life will be measure with the QLQ-MY20 questionnaire to assess the quality of life of cancer patients.
  QLQ-MY20 domain scores are averaged and transformed linearly to a score ranging from 0-100. A high score for Disease Symptoms and Side Effects of Treatment represents a high level of symptomatology or problems, whereas a high score for Future Perspective and Body Image represents better outcomes.

SECONDARY OUTCOMES:
Measure of fatigue evaluated by Piper scale | at day 0 from autograft as patient will be hospitalized.
  The Piper Fatigue Scale is composed of 22 numerically scaled, "0" to "10" items that measure four dimensions of subjective fatigue. This will give an average score that remains on the same "0" to "10"numeric scale. O is the moderate score and 10 is the worst score.
Measure of fatigue evaluated by Piper scale | at day 30 from autograft as patient will be hospitalized.
  The Piper Fatigue Scale is composed of 22 numerically scaled, "0" to "10" items that measure four dimensions of subjective fatigue. This will give an average score that remains on the same "0" to "10"numeric scale. O is the moderate score and 10 is the worst score.
Measure of fatigue evaluated by Piper scale | at day 90 from autograft as patient will be hospitalized.
  The Piper Fatigue Scale is composed of 22 numerically scaled, "0" to "10" items that measure four dimensions of subjective fatigue. This will give an average score that remains on the same "0" to "10"numeric scale. O is the moderate score and 10 is the worst score.

CONTACTS AND LOCATIONS:
Overall Officials: caroline delette, MD, Principal Investigator — CHU Amiens; Pierre Morel, MD, Principal Investigator — CHU Amiens; Fabrice Jardin, Pr, Principal Investigator — CHU Rouen; Oana Brehar, MD, Principal Investigator — CHU Rouen; Vincent Camus, MD, Principal Investigator — CHU Rouen; Nathalie Cardinael, MD, Principal Investigator — CHU Rouen; Nathalie Contentin, MD, Principal Investigator — CHU Rouen; Marie-Laure Fontoura, MD, Principal Investigator — CHU Rouen; Carole Fronville Varnier, MD, Principal Investigator — CHU Rouen; Hélène Lanic, MD, Principal Investigator — CHU Rouen; Emilie Lemasle Hue, MD, Principal Investigator — CHU Rouen; Pascal Lenain, MD, Principal Investigator — CHU Rouen; Stéphane Lepretre, MD, Principal Investigator — CHU Rouen; Anna-Lise Menard, MD, Principal Investigator — CHU Rouen; Aspasia Stamatoullas-Bastard, MD, Principal Investigator — CHU Rouen; Hervé Tilly, MD, Principal Investigator — CHU Rouen; Gandhi L Damaj, Pr, Principal Investigator — CHU CAEN; Stéphane Cheze, MD, Principal Investigator — CHU CAEN; Margaret Macro, MD, Principal Investigator — CHU CAEN
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No